CLINICAL TRIAL: NCT06544057
Title: Real-time eCounselling for Nicotine Addiction: a Feasibility Study and Pilot RCT
Brief Title: Real-time eCounselling for Nicotine Addiction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Overcome (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P-PF-03.24.0002
Record Dates: First submitted 2024-07-12; First posted 2024-08-09 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Nicotine Use Disorder
Keywords: Smoking cessation; Vaping; Public health; eHealth; Nicotine addiction; Feasibility
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Vaping

STUDY DESIGN:
Intervention Model Description: This was a two-arm Block randomised pilot trial with study centres using block randomisation comparing Wait-list and Active.
Who Masked: Outcomes Assessor
Masking Description: The blinding procedure aims to minimise bias by ensuring the outcome assessor, a member of our research team, remains unaware of participants' treatment allocation (Intervention or WLCG). This 'Single-Blind' design involves blinding the internal team's outcome assessor, who evaluates study endpoints without knowledge of participants' group assignments. To uphold blinding integrity, outcome assessors refrain from engaging with participants or study personnel. Participants and intervention administrators are not blinded due to the intervention nature
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-MI (Experimental): Behavioural Therapy (CBT) with Motivational Interviewing (MI) techniques. It comprises six individual sessions delivered via real-time video (Zoom) on mobile or computer platforms. Sessions last approximately 45 to 60 minutes each.
  Interventions: Behavioral: CBT-MI
- Wait-list (No Intervention): Control group will undergo recruitment and screening and be assigned to a wait-list, to undergo the intervention after the active group. Data collection will continue as in the active arm, to compare with that collected in the active arm

INTERVENTIONS:
Behavioral: CBT-MI — CBT-MI combines elements from Cognitive Behavioural Therapy and Motivational Interviewing in treating nicotine addiction, delivered remotely via Zoom by trained 'layperson coaches'
  Arms: CBT-MI

SUMMARY:
The goal of this clinical trial is to pilot an eHealth intervention (real-time telecounselling) in nicotine addiction. The main questions it aims to answer are:

Is the intervention likely to be efficacious in preventing an increase in Abstinence? Is the intervention likely to be efficacious in preventing an increase in nicotine consumption? Is the intervention likely to be efficacious in influencing Readiness to quit nicotine? How feasible is the intervention for developing a larger-scale trial?

Researchers will compare a range of outcome measures between the active and control arms, to see if a pilot eHealth intervention can successfully treat nicotine addiction.

DETAILED DESCRIPTION:
The goal of this clinical trial is to pilot an eHealth intervention in nicotine addiction (real-time telecounselling) . It will also attempt to better understand the psychology of nicotine addiction and craving regarding consumption behaviour. The main questions it aims to answer are:

Is the intervention likely to be efficacious in preventing an increase in Abstinence? Is the intervention likely to be efficacious in preventing an increase in nicotine consumption? Is the intervention likely to be efficacious in influencing Readiness to quit nicotine? How feasible is the intervention for developing a larger-scale trial?

Researchers will compare outcomes pre and post intervention in the active arm, and also between active and control arms, to ascertain the treatment effect of the intervention on primary (nicotine consumption, abstinence) and secondary (self-efficacy, readiness to quit, decisional balance) measures, in tests of efficacy.

Following randomisation, participants will be allocated to either the active arm or the control arm. In the active arm, participants will undergo six weekly sessions of real-time CBT-MI (Cognitive Behavioural Therapy with Motivational Interviewing), with each session lasting approximately 45 to 60 minutes. In the control arm: A Wait List Control Group (WLCG) will denote the comparator, who will undergo screening and assessment only.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-65 Years old
2. Self Reported smoking ≥ 5 cigarettes per day, or regular vaper of > 0mg nicotine
3. Desire to quit nicotine consumption
4. Willing to set a quit date
5. Able to provide written informed consent to participate -

Exclusion Criteria:

1. Enrolled in another behavioural intervention programme
2. Pregnant, breastfeeding or planning to become pregnant.
3. Individuals currently experiencing a problematic relationship with alcohol or drugs
4. Documented Cognitive Impairment
5. Individuals with a PHQ-9 score of ≥ 14 or a GAD-7 score of >12.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Abstinence status | 1 week post study: 7 days retrospective
  This is a binary indicator, suggesting whether or not participants are abstinent at point of questioning
Nicotine consumption (cigarettes, units) | Baseline; 6 weeks after the intervention
  Unit: Number of cigarettes consumed, on average, per day
Nicotine consumption (cigarettes, time) | Baseline; 6 weeks after the intervention
  Time: Time spent smoking nicotine, on average, per day
Nicotine consumption (vape, units) | Baseline; 6 weeks after the intervention
  Unit: Number of 15-minute 'episodes' of vaping, on average, per day
Nicotine consumption (vape, time) | Baseline; 6 weeks after the intervention
  Time: Time spent vaping nicotine, on average, per day

SECONDARY OUTCOMES:
Dependence and Craving (CDS) | Baseline; 6 weeks after the intervention
  Cigarette dependence and craving experiences will be assessed using the Cigarette Dependence Scale (CDS), which measures various aspects of nicotine dependence, including withdrawal symptoms, desire to quit, time spent using, and the effects of consumption on activities. The scale has possible values of 1, 2, 3, 4, 5. On this ordinal scale, higher values denote stronger agreement.
Dependence and Craving (EDS) | Baseline; 6 weeks after the intervention
  The (Electronic) e-Cigarette Dependence Scale (EDS) captures similar dimensions of dependence specific to e-cigarette use and will be administered at the same time points as the Cigarette Dependence Scale (CDS), which measures various aspects of nicotine dependence, including withdrawal symptoms, desire to quit, time spent using, and the effects of consumption on activities. This scale measures the level of nicotine dependence in those who use e-cigarettes or vapes. The scale has possible values of 1, 2, 3, 4, 5. On this ordinal scale, higher values denote stronger agreement.
Readiness to Quit | Baseline; Every week during the intervention
  Participants' readiness to quit smoking will be assessed using the contemplation ladder (CL), which measures their current stage of change in the quitting process. The Contemplation Ladder (CL) measures readiness to quit using an 11-point Likert scale, ranging from "No thoughts of quitting" (0) to "Taking action to quit" (10). he possible values of the measure were 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11. On this ordinal scale, higher values denote stronger agreement regarding readiness to quit.
Perceived Smoking Abstinence Efficacy as assessed by questionnaire measuring participants' confidence in their ability to quit smoking, and their resistance to temptation to relapse | Baseline; Every week during the intervention
  The questionnaire comprises items related to positive social situations, negative affect situations, and habitual/craving situations. Responses will be recorded on a 5-point Likert scale ranging from 'Not at all tempted' to 'Extremely tempted'. The possible values of the measure were 1, 2, 3, 4, 5, 6, 7, 8, 9. On this ordinal scale, higher values denote stronger agreement regarding self-efficacy in nicotine abstinence.
Decisional balance | Baseline; Every week during the intervention
  'Decisional balance' evaluates the pros and cons of nicotine consumption and quitting. This scale measures participant's relative weighing of the pros and cons of smoking/vaping. The possible values of the measure were 1, 2, 3, 4, 5. On this ordinal scale, higher values denote stronger agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Hayward, BSc, Study Director — Overcome
Locations (1):
- Key contact, Leicester, Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No
A member of the research team (HH) will regularly monitor the trial and its delivery to ensure ongoing study protocol compliance. In the event of deviations from the study protocol or unexpected events, the study team will promptly document and report such occurrences to the designated individuals and the Institutional Ethics review board, following the established reporting timelines. All study-related documentation, including data collection forms and interview transcripts, will be securely stored in password-protected electronic databases, adhering to data security and confidentiality guidelines.

REFERENCES:
- [Background] Biener L, Abrams DB. The Contemplation Ladder: validation of a measure of readiness to consider smoking cessation. Health Psychol. 1991;10(5):360-5. doi: 10.1037//0278-6133.10.5.360. PMID 1935872
- [Background] Etter JF, Le Houezec J, Perneger TV. A self-administered questionnaire to measure dependence on cigarettes: the cigarette dependence scale. Neuropsychopharmacology. 2003 Feb;28(2):359-70. doi: 10.1038/sj.npp.1300030. PMID 12589389
- [Background] Morean ME, Krishnan-Sarin S, Sussman S, Foulds J, Fishbein H, Grana R, O'Malley SS. Psychometric Evaluation of the E-cigarette Dependence Scale. Nicotine Tob Res. 2019 Oct 26;21(11):1556-1564. doi: 10.1093/ntr/ntx271. PMID 29301008
- [Background] Prochaska JO, Velicer WF. The transtheoretical model of health behavior change. Am J Health Promot. 1997 Sep-Oct;12(1):38-48. doi: 10.4278/0890-1171-12.1.38. PMID 10170434
- [Background] Abrams, D. B., Herzog, T. A., Emmons, K. M., Linnan, L., & Stages of Change Working Group. (2000). Predicting smoking cessation from intentions and plans: Does type of smoker matter? Health Psychology, 19(1S), 24-33. DOI: 10.1016/j.addicn.2023.100068.
- [Background] Fidancı, I., Sümer, H. C., & Fırat, S. (2017). The role of emotion regulation difficulties and smoking-related cognitions in understanding anxiety and smoking among treatment-seeking smokers. Journal of Cognitive Psychotherapy, 31(3), 227-240
- [Background] Velicer WF, Diclemente CC, Rossi JS, Prochaska JO. Relapse situations and self-efficacy: an integrative model. Addict Behav. 1990;15(3):271-83. doi: 10.1016/0306-4603(90)90070-e. PMID 2378287

DOCUMENTS (1):
  • Informed Consent Form (2024-07-11): https://cdn.clinicaltrials.gov/large-docs/57/NCT06544057/ICF_000.pdf